CLINICAL TRIAL: NCT05606315
Title: RemImazolam Besylate for ICU-sedation in Patients With Mechanical Ventilation After Oral and Maxillofacial Surgery: Multicenter, Randomized, Non-inferiority Clinical Study
Brief Title: RemImazolam Besylate for ICU-sedation in Patients With Mechanical Ventilation After Oral and Maxillofacial Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-341
Record Dates: First submitted 2022-11-02; First posted 2022-11-04 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Remimazolam Besylate; Sedation; ICU
Keywords: Remimazolam besylate; Oral cancer; Sedation; ICU
MeSH Terms: conditions — Mouth Neoplasms | interventions — Propofol; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam besylate (Experimental): Remimazolam besylate is a new ultra-short-acting benzodiazepine drug, which is a benzodiazepine central nervous system inhibitor. It can bind to central GABAA receptors and produce sedative effects in animal experiments. Currently, it is used in painless diagnosis and treatment sedation, colonoscopy sedation, general anesthesia, ICU sedation and local anesthesia sedation.
  Interventions: Drug: Remimazolam Besylate
- propofol (Active Comparator): Propofol, known chemically as 2, 6-diisopropyl phenol, is an organic compound with the chemical formula C12H18O and is a short-acting intravenous anesthetic used for the induction and maintenance of general anesthesia. It is often used in conjunction with epidural or spinal anesthesia, as well as with analgesics, muscle relaxants, and inhalation anesthetics.
  Interventions: Drug: Propofol
- midazolam (Active Comparator): Midazolam, an organic compound with the chemical formula C18H13ClFN3, is used clinically to treat insomnia and can also be used to induce sleep during surgery or diagnostic tests.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam Besylate — NS 50ML + Remimazolam besylate(50mg , 2mg:2ml), IV-Pump,maintenance dose 0.5-3mg/kg/h.
  Arms: Remimazolam besylate
Drug: Propofol — Propofol (50ml, 0.5g), IV-Pump, maintenance dose 0.3-4.0mg/kg/h.
  Arms: propofol
Drug: Midazolam — Midazolam (10mg,2ml), IV-Pump, maintenance dose 0.02-0.1mg/kg/h.
  Arms: midazolam

SUMMARY:
Remimazolam besylate, as a new benzodiazepine drug, showing rapid clearance and moderate distribution of pharmacokinetic changes. The study will further explore the safety and effectiveness of remimazolam besylate n the sedation of mechanically ventilated patients after oral and maxillofacial surgery in the ICU.

DETAILED DESCRIPTION:
Remimazolam besylate is a new type of ultra-short-acting benzodiazepine, showing rapid clearance and moderate distribution of pharmacokinetic changes. Remimazolam has been widely studied for programmed sedation in endoscopic procedures such as gastroenteroscopy and bronchoscopy. Remimazolam, as a short-acting sedative agent that is not metabolized by liver or kidney, can achieve rapid and reversible sedation and has the potential to shorten the duration of mechanical ventilation.

In the oral and maxillofacial surgical treatment, the use of microvascular free tissue transfer for reconstruction is one of the common operations. In order to avoid mechanical damage to the transplanted reconstructed tissue due to spontaneous movement, patients undergoing major head and neck reconstruction surgery are considered to require postoperative deep sedation for a certain period of time (RASS score required -4/-5 points). Deep sedation may cause hypotension and lead to reduced flap perfusion pressure, increasing the risk of hypoperfusion and flap necrosis, thus requiring close postoperative monitoring in the ICU.

Therefore, there is an urgent need for a sedative drug that can achieve rapid and sufficient sedation, does not inhibit breathing and can reduce the amount of patients or rapid recovery after drug withdrawal without increasing delirium. Based on the deficiencies of currently used sedatives and the potential advantages of remimazolam, we hypothesize that remimazolam can shorten the extubation time and lower the adverse reaction rate in patients with oropharyngeal cancer after mechanical ventilation sedation.

This clinical study was a randomized, multi-center, parallel-controlled, non-inferior clinical study. After signing the informed consent, participants meeting the inclusion/exclusion criteria will be randomly assigned to the treatment group (ramazolam besylate) and the control group (propofol, midazolam) in a ratio of 1:1:1, with a total of 285 participants recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* After undergoing oral and maxillofacial surgery, it is expected that a ventilator will be needed to assist with breathing;
* mechanical ventilation patients with expected ICU stay time <72h;
* People who need immediate sedative treatment;
* Obtain informed consent from subject or legal representative;

Exclusion Criteria:

* Pregnancy；
* Can not get RASS score from patients;
* Allergy to drugs;
* Proven acute and severe intracranial or spinal nerve disease due to vascular, infection, intracranial dilation, or injury;
* Uncompensated acute circulatory failure at randomization (severe hypotension with MAP<50 mmHg despite adequate fluid resuscitation and vasopressor therapy);
* Severe bradycardia (heart rate <50 beats/min) or degree II-III heart block (unless a pacemaker is installed);
* A history of long-term use of benzodiazepines or opioids;
* Subjects receiving sedation for indications other than to tolerate ventilators (e.g., epilepsy);
* Continuous sedation is unlikely to be required during mechanical ventilation (e.g. Guillain-Barre syndrome);
* Patients determined by the clinician to be unlikely to be removed from mechanical ventilation, such as diseases/injuries that primarily affect respirator neuromuscular function and conditions that clearly require long-term ventilation support (such as high spinal cord injury);
* Participation in any other interventional study (any study that assigns subjects to different treatment groups and/or performs unconventional diagnostic or monitoring procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Extubation time | From date of using the intervention drugs until the date of extubation, up to 28 days.
  The time from discontinuation of sedation to withdrawal of tracheal catheter.

SECONDARY OUTCOMES:
Time to recovery | From date of using the intervention drugs until the date of recovery, up to 28 days.
  The time from withdrawal of sedation to recovery.
Drug onset time | From date of using the intervention drugs until the date of recovery, up to 28 days.
  The time from discontinuation of sedation to meeting the sedation score requirements (RASS score < -3).
Time to reach the required sedation score | From date of using the intervention drugs until the date of recovery, up to 28 days.
  The proportion of time spent meeting sedation requirements (RASS score <-3) to total time spent on medication
Mechanical ventilation time during ICU | From the time you enter ICU to the time you leave ICU.
  Time from insertion to withdrawal of tracheal catheter.
Length of ICU stay and total hospital stay | From hospitalization to discharge.
  Time from admission to ICU to leave ICU;The time from admission to discharge.
Adverse event rate | From date of using the intervention drugs until the date of leaving hospital.
  The proportion of cases with adverse events to the total number of cases for evaluation of adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Southern medical university Nanfang hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong